CLINICAL TRIAL: NCT05450835
Title: Comparison Of Short-term Outcomes Between OGT-assisted Overlap Esophagojejunostomy And Traditional Overlap Method In Patients With Siewert III/II Esophagogastric Junction Cancer Or Gastric Cancer
Brief Title: OGT-assisted Overlap Esophagojejunostomy Versus Traditional Overlap Method
Acronym: OGT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-202
Record Dates: First submitted 2022-07-01; First posted 2022-07-11 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Gastric Cancer
Keywords: Gastric/gastroesophageal junction (G/GEJ) tumors; Laparoscopy total gastrectomy; Overlap esophagojejunostomy; OGT
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: In OGT group,the oesophagojejunostomy was performed with OGT-assisted overlap method.
  In overlap group, the oesophagojejunostomy was performed as reported by Inaba et al.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): In OGT group,After the enterotomy was made, the nasogastric tube was pulled out 3 cm from the oesophagal lumen to connect with the OGT. Next, the anvil fork sleeved with OGT insert into the oesophageal mucosa canal by movement of the connection of fork -OGT -gastric tube. Then, the anaesthesiologist continued to pull back the nasogastric tube for 10 cm to ensure that the stapler would not clamp the nasogastric tube. After that, the surgeon began to fire the stapler to perform side-to-side esophagojejunostomy.
  Interventions: Procedure: OGT group
- Arm B (Active Comparator): In overlap group, the oesophagojejunostomy was performed as reported by Inaba et al. After firing the stapler, two openings were converted into a single entry hole to create an end-to-side oesophagojejunostomy, and the entry hole was closed with full-thickness running suture using barbed sutures intracorporeally.
  Interventions: Procedure: Overlap group

INTERVENTIONS:
Procedure: OGT group — In OGT group,the nasogastric tube was pulled out 3 cm from the oesophagal lumen to connect with the OGT. Meanwhile, the OGT was sleeved on anvil fork extracorporeally and the linear stapler was put into abdomen through trocar on the right side and then cartridge fork was inserted through jejunum opening towards the oral side of the lumen. Next, the anvil fork sleeved with OGT insert into the oesophageal mucosa canal by movement of the connection of fork -OGT -gastric tube.
  Arms: Arm A
Procedure: Overlap group — In overlap group, the oesophagojejunostomy was performed as reported by Inaba et al.
  Arms: Arm B

SUMMARY:
Abstract Background Our previous studies have shown OGT method significantly simplified overlap esophagojejunostomy with good short-term outcomes, and provided new perspectives for optimizing esophagojejunostomy. However, the safety and efficiency of OGT method still need evidence of randomized controlled trial.

Methods: This trial is a prospective, multicenter, randomized, controlled, open, and superiority trial. Three hundred and forty-four patients who met the inclusion criteria and did not accord with the exclusion criteria will be randomly divided into OGT group(n=172) and traditional group(n=172). The primary purpose of this study is to evaluate time of oesophagojejunostomy of OGT method compared with traditional method for Siewert III/II esophagogastric junction cancer and gastric cancer. The second purpose is to evaluate the success rate of inserting anvil fork into esophageal lumen at first attempt, attempts of inserting anvil fork into esophagus, early postoperative complications,recovery course and compare the postoperative hospital stay of the patients enrolled in this study.

Discussion: This trial is the first prospective randomized two-arm controlled study to determine the safety and efficiency of OGT method compared with traditional overlap method. Through this trial, we hope to show that experienced surgeons can safely perform OGT-assisted overlap esophagojejunostomy for Siewert III/II esophagogastric junction cancer and gastric cancer.

DETAILED DESCRIPTION:
Methods Objectives This trial is a prospective, multicenter trial for OGT-assisted overlap esophagojejunostomy and traditional overlap method during totally laparoscopic total gastrectomy for Siewert III/II esophagogastric junction cancer and gastric cancer. The primary purpose of this study is to evaluate the time of oesophagojejunostomy of OGT method compared with traditional overlap method for Siewert III/II esophagogastric junction cancer and gastric cancer. The second purpose is to evaluate the success rate of inserting anvil fork into esophageal lumen at first attempt, attempts of inserting anvil fork into esophagus, early postoperative complications,recovery course and compare the postoperative hospital stay of the patients enrolled in this study.

Study design This trial is a prospective, multicenter, randomized, controlled, open, and superiority trial comparing the safety of OGT method during TLTG for Siewert III /II esophagogastric junction cancer and gastric cancer compared with traditional overlap method .

Participating surgeons To participate in this trial, the responsible surgeons should meet the following qualifications: first, completing at least 50 cases of TLTG with D2 lymphadenectomy;second, passing the blind review of surgery video. Briefly, the applicants should provide the videos of TLTG with traditional overlap and OGT method in recent 3 months (three cases each) to the CLASS Research Council.CLASS Research Council will select two videos of traditional overlap and OGT method separately, and randomly appoint three experts to peer review blindly. When three experts unanimously approved it, the applicant will be permitted to participate in this study as a researcher.

Sample size calculation This is a superiority verification study on clinical efficiency, with the time of oesophagojejunostomy as the main index for efficiency evaluation. Our center's early OGT Overlap esophagojejunal anastomosis takes only 21 minutes, compared to 30-32 minutes for the conventional technique. The experimental group has a mean standard deviation of 6, while the control group has a mean standard deviation of 8. The ratio of the two groups is 1:1, and the superiority threshold is set at 7. With a one-sided error of 0.05 and a power test of 0.8, we calculated the required sample size for each group as 156 cases. Given a maximum dropout rate of about 10%, the final sample size for each group was set at 172 cases, totaling 344 cases.

Inclusion criteria Aged 18-75 years; Primary lesion is pathologically diagnosed as gastric adenocarcinoma; Expected to live more than 1 year; Tumor located located in gastroesophageal junction (GEJ) involve esophagus no more than 2cm, or in the upper, upper to middle, or entire stomach, and intend to perform laparoscopic total gastrectomy with D2 lymphadenectomy No history of upper abdominal surgery (except for laparoscopic cholecystectomy); Preoperative performance status (ECOG, Eastern Cooperative Oncology Group) of 0 or 1; Preoperative ASA (American Society of Anesthesiologists) scoring: I-III; Sufficient organ functions; Written informed consent.

Exclusion criteria Women during pregnancy or breast-feeding; Body temperature ≥ 38 °C before surgery or infectious disease with a systemic therapy indicated; Severe mental disease; Confirmed stage IV (AJCC 8th) during surgery Severe respiratory disease; Severe hepatic and renal dysfunction; Unstable angina pectoris or history of myocardial infarction within 6 months; History of cerebral infarction or cerebral hemorrhage within 6 months; Gastric cancer complications (bleeding, perforation, obstruction) that requiring emergency surgery.

Randomized grouping In this study, the central dynamic, stratified randomization method is adopted, and the factors including age, TNM stage, tumor location, neoadjuvant, BMI, and investigators, are considered. After each case is enrolled, the research center will arrange the research assistant to send the information of included cases (age,TNM stage, tumor location, neoadjuvant, and BMI) to the data center. After analyzing the case information by the center randomization department, the case grouping will be determined.

Quality control To ensure the rationality of the ESJ procedure, a series of photographs of ESJ (traditional and OGT) are taken for assessment. All photographs will be saved and submitted to CLASS data center within 1 week after the operation. The CLASS Research Committee will monitor and review regularly to ensure the quality of operation.

Outcome measurements

Primary endpoint:

Time of oesophagojejunostomy: time starts from making the entry hole for the anastomosis on the oesophagealstump, to the end of the common entry hole was closed using barbed threads.

The secondary endpoint of this study is early postoperative complications, the success rate of inserting anvil fork into oesophagal lumen at first attempt, the number of attempts to insert anvil fork into oesophagus and postoperative recovery course, which is assessed by time to first ambulation, flatus, liquid diet, soft diet, etc. In addition, the length of postoperative hospital stay will be recorded.

Follow-up The patients in both groups will be followed up 6 months after operation. A physical examination, a complete blood count, blood biochemical examination (albumin, prealbumin, total bilirubin, direct bilirubin, AST, ALT, creatinine, blood urea nitrogen, and blood glucose), and serum tumor markers (AFP, CEA, CA19-9, CA12-5, and CA72-4) analyses will be performed. In addition, imageological examination (total abdominal and pelvic enhanced CT, chest X-ray, upper gastrointestinal tract iodine imaging, gastroscopy, ultrasonography, whole body bone scan, PET-CT, etc.) will also be performed if needed. All the results will be recorded and evaluated by the specialist.

Statistical analysis Statistical analysis will be performed with SPSS 25.0 (SPSS Inc., Chicago, IL, USA). Continuous variables with normal distribution are expressed as the mean ± standard deviation, and continuous variables with a skewed distribution are expressed as the median (interquartile range [IQR]) and were compared across groups using. Continuous variables were compared across groups using the independent t-test or Mann-Whitney U test if the data were highly skewed. Categorical variables are expressed as the number and percentage and were compared with the chi-square test or Fisher's exact test(if a variable's exact theory frequency was less than 1). P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years;
* Primary lesion is pathologically diagnosed as gastric adenocarcinoma;
* Expected to live more than 1 year;
* Tumor located located in gastroesophageal junction (GEJ) involve esophagus no more than 2cm, or in the upper, upper to middle, or entire stomach, and intend to perform laparoscopic total gastrectomy with D2 lymphadenectomy
* No history of upper abdominal surgery (except for laparoscopic cholecystectomy);
* Preoperative performance status (ECOG, Eastern Cooperative Oncology Group) of 0 or 1;
* Preoperative ASA (American Society of Anesthesiologists) scoring: I-III;
* Without preoperative radiotherapy;
* Did not found metastasis preoperatively and intraoperatively;
* Sufficient organ functions;
* Written informed consent.

Exclusion Criteria:

* Women during pregnancy or breast-feeding;
* Body temperature ≥ 38 °C before surgery or infectious disease with a systemic therapy indicated;
* Severe mental disease;
* Confirmed stage IV (AJCC 8th) during surgery
* Severe respiratory disease;
* Severe hepatic and renal dysfunction;
* Unstable angina pectoris or history of myocardial infarction within 6 months;
* History of cerebral infarction or cerebral hemorrhage within 6 months;
* Gastric cancer complications (bleeding, perforation, obstruction) that requiring emergency surgery;
* Performing hyperthermic intraperitoneal chemotherapy (HIPEC) after surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Time of oesophagojejunostomy | 1 Days
  Time starts from making the entry hole for the anastomosis on the oesophagealstump, to the end of the common entry hole was closed using barbed threads.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Yu, Ph.D, Principal Investigator — Nanfang Hospital, Southern Medical University; Quan Wang, Ph.D, Principal Investigator — The First Hospital of Jilin University; Kai Ye, Ph.D, Principal Investigator — Fujian Medical University 2nd Affiliated Hoapital; Chuanfa Fang, Ph.D, Principal Investigator — Ganzhou City People Hospital; Feirang Zhang, Ph.D, Principal Investigator — First Affiliated Hospital of Shantou University Medical College; Wei Wang, Ph.D, Principal Investigator — The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine; Wenqing Hu, Ph.D, Principal Investigator — The People's Hospital of Changzhi; Junjiang Wang, Ph.D, Principal Investigator — Guangdong Provincial People's Hospital; Lei Lian, Ph.D, Principal Investigator — Sixth affiliated hospital of Sun Yat-sen University; Jiaquan Zhu, Ph.D, Principal Investigator — First Hospital of China Medical University; Yi Zhang, Ph.D, Principal Investigator — The Third Xiangya Hospital of Central South University; Shuai Xiao, Ph.D, Principal Investigator — The First Affiliated Hospital of Nanhua University
Locations (12):
- China (12):
  - Fujian Medical University 2nd Affiliated Hoapital, Quanzhou, Fujian
  - Nanfang Hospital, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sixth affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Ganzhou City People Hospital, Ganzhou, Guangxi
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanhua University, Hengyang, Hunan
  - The First Hospital Of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The People's Hospital of Changzhi, Changzhi, Shanxi

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available for the investigation.
Supporting Information: Study Protocol, SAP
Time Frame: August, 2022-August, 2025
Access Criteria: All the accession for research will be admitted.